CLINICAL TRIAL: NCT03212170
Title: [18F]Fluorofuranylnorprogesterone (FFNP) PET/MR Imaging of Progesterone Receptor Expression in Invasive Breast Cancer
Brief Title: FFNP-PET/MR Imaging of Progesterone Receptor Expression in Invasive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-0533; UW17034 / UW23007 (Other: UWCCC ID); A539300 (Other: UW Madison); SMPH\RADIOLOGY\RADIOLOGY (Other: UW Madison); 4UL1TR000427-10 (NIH); 1UL1TR002373-01 (NIH); Protocol Version 11/2/2022 (Other: UW Madison)
Record Dates: First submitted 2017-06-30; First posted 2017-07-11 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Invasive Breast Cancer
Keywords: Invasive Breast Cancer; Metastatic Breast Cancer; PR Positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FFNP PET/MRI (Experimental): 18F-Fluorofuranylnorprogesterone (FFNP) administration for PET/MRI imaging to assess biopsy-proven primary PR+ breast malignancies.
  Interventions: Drug: [18F]Fluorofuranylnorprogesterone (FFNP) PET/MR Imaging

INTERVENTIONS:
Drug: [18F]Fluorofuranylnorprogesterone (FFNP) PET/MR Imaging — 18F-Fluorofuranylnorprogesterone (FFNP) PET/MR Imaging tracer
  Other Names: FFNP

SUMMARY:
The goal of this research is to test the accuracy of PET/MRI imaging with 18F-fluorofuranylnorprogesterone (FFNP) for measuring progesterone receptor (PR) expression in patients with invasive breast cancer. The hypothesis is that FFNP SUVmax from PET/MRI will correlate well against the semi-quantitative PR immunohistochemistry score.

DETAILED DESCRIPTION:
Integrated whole-body magnetic resonance imaging (MRI)-positron emission tomography (PET) scanners have recently been introduced for clinical use. This technology combines the anatomic and perfusion data obtained with dynamic contrast enhanced (DCE) MRI with functional imaging data obtained from PET. For breast imaging, the combination of MRI and PET has important potential to improve diagnostic accuracy and provide molecular characterization of breast cancer. The overall purpose of this research is to test the accuracy of PET/MRI imaging with 18F-fluorofuranylnorprogesterone (FFNP) for measuring progesterone receptor (PR) expression in patients with invasive breast cancer.

This is a prospective, one-arm, study which will enroll patients with newly diagnosed breast cancer scheduled for diagnostic breast MRI for preoperative staging/extent of disease evaluation as part of standard of care. Participation in this research study includes a directed breast PET/MRI with the investigational radiopharmaceutical, FFNP. FFNP uptake of the known, biopsy-proven malignancy will be measured on the PET/MRI examinations using standardized uptake values (SUV) and tumor-to-normal tissue ratios.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older
* Diagnosis of biopsy-proven invasive breast cancer measuring at least 1.0 cm in diameter by any imaging modality
* Biopsy-proven PR-positive or PR-negative invasive breast cancer
* Undergoing diagnostic breast MRI ordered by the referring clinician for staging and extent of disease

Exclusion Criteria:

* Inability or unwillingness to provide informed consent to the study
* Participants currently undergoing neoadjuvant chemotherapy/endocrine therapy or those who have received chemotherapy/endocrine therapy within 6 months prior to the MRI
* Participants who have had neoadjuvant chemotherapy/endocrine therapy, surgical intervention, or radiation for the current biopsy-proven malignancy
* Participants with breast expanders
* Participants who are or might be pregnant or lactating
* Participants with a contraindication to gadolinium based contrast agents, including allergy or impaired renal function (per University of Wisconsin Health Guidelines)
* Participants with a history of allergic reaction attributable to compounds of similar chemical or biologic composition to FFNP
* Participants in liver failure as judged by the patient's physician
* Participants with standard contraindications to MRI, including claustrophobia and metallic implants incompatible with MRI
* Participants requiring intravenous (IV) conscious sedation for imaging are not eligible; participants requiring mild, oral anxiolytics for the clinical MRI will be allowed to participate as long as the following criteria are met:

  * The subject has their own prescription for the medication
  * The informed consent process is conducted prior to the self-administration of this medication
  * They come to the research visit with a driver
* Participants unable to lie prone for 30 minutes for imaging

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women are being targeted for this research as breast MRI is not utilized for male breast cancer patients which comprises only 1% of all breast cancer cases.
Enrollment: 21 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Fowler, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from December 2017 to November 2024.
Groups:
- FFNP PET/MRI: 18F-Fluorofuranylnorprogesterone (FFNP) administration for Positron Emission Tomography / Magnetic Resonance Imaging (PET/MRI) to assess biopsy-proven primary PR+ breast malignancies.
  [18F]Fluorofuranylnorprogesterone (FFNP) PET/MR Imaging: 18F-Fluorofuranylnorprogesterone (FFNP) PET/MR Imaging tracer
Period: Overall Study
Arm/Group | FFNP PET/MRI
Started | 21
Analysis Population | 20
Completed | 20
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | FFNP PET/MRI
Number analyzed (Participants) | 21
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 1
  40-49 years | 3
  50-59 years | 12
  60-69 years | 4
  70-79 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Correlation Coefficient Between FFNP Uptake and Allred Score
Description: To compare FFNP uptake of biopsy-proven primary PR+ breast malignancies measured using PET/MRI with the reference standard of PR immunohistochemistry (IHC) using a semi-quantitative score obtained by using the Allred score (0-8; the higher the score, the more receptors were found). The correlation of the two measures will be evaluated with Pearson's correlation coefficient. The null hypothesis is H0: p0=0.50 and the alternative hypothesis is H1: p1 =0.75.
Time Frame: Up to 1 day
Measure: Number; unit: correlation coefficient (rho)
Arm/Group | FFNP PET/MRI
Number analyzed (Participants) | 20
correlation coefficient (rho) | 0.3215
Statistical Analysis 1: Comparison: FFNP PET/MRI; Test type: Other — Pearson correlation statistical test; p = 0.1347, two-sided hypothesis test

2. Secondary Outcome: Test-Retest Reproducibility
Description: Tumor uptake of FFNP and the ability to reproduce this measure, will be quantified in the 5 subjects who elect to undergo a second imaging session, using summary statistics of tumor FFNP uptake for each reading for PET/MRI. The analysis will be done separately for each reader.
Time Frame: Up to 4 weeks
Population: test-retest completed on a subset of the population, only 1 participant volunteered
Measure: Mean (Standard Deviation); unit: SUVmax
Groups:
- FFNP PET/MRI (Re-test): 18F-Fluorofuranylnorprogesterone (FFNP) administration for PET/MRI imaging to assess biopsy-proven primary PR+ breast malignancies.
Arm/Group | FFNP PET/MRI | FFNP PET/MRI (Re-test)
Number analyzed (Participants) | 1 | 1
SUVmax | NA (NA) — Only 1 participant volunteered, data is insufficient to analyze test-retest reproducibility. | NA (NA) — Only 1 participant volunteered, data is insufficient to analyze test-retest reproducibility.

3. Secondary Outcome: Intra and Inter-Observer Assessment
Description: The variability of observer assessment of tumor FFNP uptake will be measured. The intra- and inter-reader agreement of SUV values for tumor FFNP uptake will be analyzed with Bland-Altman plots and 95% limits of agreement. Analyses will be conducted on a per-lesion basis, and repeat tumors within the same patient will be assumed to be independent.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: SUVmax
Groups:
- FFNP PET/MRI (Reader 1 Assessment): 18F-Fluorofuranylnorprogesterone (FFNP) administration for PET/MRI imaging to assess biopsy-proven primary PR+ breast malignancies.
  [18F]Fluorofuranylnorprogesterone (FFNP) PET/MR Imaging: 18F-Fluorofuranylnorprogesterone (FFNP) PET/MR Imaging tracer
- FFNP PET/MRI (Reader 2 Assessment): 18F-Fluorofuranylnorprogesterone (FFNP) administration for PET/MRI imaging to assess biopsy-proven primary PR+ breast malignancies.
Arm/Group | FFNP PET/MRI (Reader 1 Assessment) | FFNP PET/MRI (Reader 2 Assessment)
Number analyzed (Participants) | 20 | 20
SUVmax | 2.76 (1.536) | 2.629 (1.568)
Statistical Analysis 1: Comparison: FFNP PET/MRI (Reader 1 Assessment) vs FFNP PET/MRI (Reader 2 Assessment); Test type: Other — Bland-Altman statistical test; Mean Difference (Final Values) = 0.1308, 95% CI 2-sided [-0.282 to 0.544]

4. Secondary Outcome: Correlation Coefficient Between Tumor FFNP Uptake With Oncotype DX Score
Description: Estimate the association of tumor FFNP uptake (continuous SUVmax) with research-based Oncotype DX scores (0-100). The risk score (0-100) is generated from expression levels of sixteen cancer related genes and five reference genes. Scores are further categorized as low-risk (0-17), intermediate-risk (18-30), and high-risk (31-100). Pearson's or Spearman's rank correlation will be used to evaluate the association between FFNP uptake and research-based Oncotype DX score. The correlation coefficient (rho) and 95% confidence interval will be reported.
Time Frame: Up to 4 weeks
Measure: Number (95% Confidence Interval); unit: correlation coefficient (rho)
Arm/Group | FFNP PET/MRI
Number analyzed (Participants) | 20
correlation coefficient (rho) | -0.377 [-0.797 to 0.2873]
Statistical Analysis 1: Comparison: FFNP PET/MRI; Test type: Other; p = 0.2521, Pearson Correlation Statistical Test

5. Secondary Outcome: Distinguishing Between PR Negative and PR Positive Breast Cancer Reported as Area Under the Curve (AUC)
Description: To evaluate the optimal cut-point of FFNP uptake for distinguishing between PR-negative and PR-positive invasive breast cancer. Receiver operating characteristic (ROC) curve analysis will be performed to determine the optimal cut-point for FFNP uptake to distinguish PR-positive from PR-negative invasive breast cancer, as defined by the clinical pathology report. The AUC for the ROCs and their respective two-sided 95% confidence intervals will be calculated using logistic regression. The optimal cut-off point will be determined by considering the FFNP uptake value with the maximum sensitivity and specificity. The analysis will be done separately for each reader, AUC is reported here.
Time Frame: up to 4 weeks
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | FFNP PET/MRI (Reader 1 Assessment) | FFNP PET/MRI (Reader 2 Assessment)
Number analyzed (Participants) | 20 | 20
probability | 0.80 [0.361 to 0.99] | 0.70 [0.47 to 0.93]

6. Secondary Outcome: Distinguishing Between PR Negative and PR Positive Breast Cancer Reported as Optimal Cut Point
Description: To evaluate the optimal cut-point of FFNP uptake for distinguishing between PR-negative and PR-positive invasive breast cancer. Receiver operating characteristic (ROC) curve analysis will be performed to determine the optimal cut-point for FFNP uptake to distinguish PR-positive from PR-negative invasive breast cancer, as defined by the clinical pathology report. The AUC for the ROCs and their respective two-sided 95% confidence intervals will be calculated using logistic regression. The optimal cut-off point will be determined by considering the FFNP uptake value with the maximum sensitivity and specificity. The analysis will be done separately for each reader, optimal cut point is reported here.
Time Frame: up to 4 weeks
Measure: Number; unit: SUVmax
Arm/Group | FFNP PET/MRI (Reader 1 Assessment) | FFNP PET/MRI (Reader 2 Assessment)
Number analyzed (Participants) | 20 | 20
SUVmax | 1.96 | 1.96

ADVERSE EVENTS:
Time Frame: up to 24 hours
Description: Adverse events occurring within 24 hours after FFNP infusion will be recorded by the study coordinator who will contact the subject within 1 to 3 days after FFNP administration.
Arm/Group | FFNP PET/MRI
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FFNP PET/MRI (N=20)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT03212170/Prot_SAP_000.pdf